CLINICAL TRIAL: NCT03023995
Title: Coronally Advanced Flap With Connective Tissue Graft and PRF for Recession Coverage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. D. Y. Patil Dental College & Hospital (Other)
Responsible Party: Principal Investigator, Santosh Martande, Lecturer, Dr. D. Y. Patil Dental College & Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DYP/2010/2PE
Record Dates: First submitted 2017-01-11; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAF with Platelet Rich Fibrin (Experimental): In test group, preparation of PRF was carried out, after which the flap was coronally positioned over the membrane to completely cover it.
  Interventions: Procedure: CAF with Platelet rich fibrin
- CAF with connective tissue graft (Active Comparator): In control group, connective tissue graft harvesting was carried out which was followed by placement of connective tissue graft on the recipient site. The connective tissue graft was placed on the recipient site and secured in position with 5-0 vicryl sutures
  Interventions: Procedure: CAF with connective tissue graft

INTERVENTIONS:
Procedure: CAF with Platelet rich fibrin — In test group, preparation of PRF was carried out, after which the flap was coronally positioned over the membrane to completely cover it and secured with 4-0 non resorbable sutures.
  Arms: CAF with Platelet Rich Fibrin
Procedure: CAF with connective tissue graft — In control group, connective tissue graft was harvested, after which the flap was coronally positioned over the graft to completely cover it and secured with 4-0 non resorbable.
  Arms: CAF with connective tissue graft

SUMMARY:
Over the years, numerous surgical techniques such as free autografts and pedicle grafts have been introduced to correct gingival recession defects. Combination grafts with either autografts or allografts, and newer concepts of guided tissue regeneration (GTR), platelet concentrates, etc., were developed more recently to correct mucogingival defects. The use of PRF in various surgical procedures such as degree II furcations, intrabony defects, sinus floor segmentation during implant placement and on facial plastic surgeries have shown promising results. However to our knowledge, till this study was completed, no studies have been reported with the clinical outcomes of autologous platelet rich fibrin membrane for the treatment of localized gingival recession defects.

Hence, this study was designed to compare coronally advanced flap with platelet rich fibrin membrane versus subepithelial connective tissue graft in treatment of Miller's Class I and Class II gingival recession defects.

DETAILED DESCRIPTION:
The study design consist of twenty sites from ten patients were randomly selected by tossing the coin for the study, which are divided into test group( Root coverage was performed by coronally advanced flap with platelet rich fibrin membrane) and Control group (Root coverage was performed with coronal advanced flap with subepithelial connective tissue graft.)

The Surgical Procedure consist of i) Preparation of the recipient bed: After adequate anesthesia, trapezoidal flap was designed using three incisions which is followed by reflection of partial thickness flap was raised apical to the crest of the osseous dehiscence. A periosteal releasing incision was given to enable the coronal advancement of the flap. Following this, root planing was done and the mesial and distal interdental papillae were deepithelialized.

The exposed root surface was conditioned with tetracycline hydrochloride for four mins. (The tetracycline hydrochloride powder was mixed with saline in dappen dish and then applied on the root surface).

In test group, preparation of PRF was carried out, after which the flap was coronally positioned over the membrane to completely cover it and secured with non resorbable sutures. The surgical area was covered with a non - eugenol periodontal dressing with post-operative antibiotics and analgesics and post-operative instructions that were given to all the patients.

In control group, connective tissue graft harvesting was carried out which was followed by placement of connective tissue graft on the recipient site. The connective tissue graft was placed on the recipient site and secured in position with vicryl sutures. The flap was coronally positioned over the connective tissue graft and secured with non resorbable sutures. The recipient bed was covered with a non-eugenol periodontal dressing with post-operative antibiotics and analgesics and post- operative instructions that were given to all the patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with age group between 20 to 55 years,
* Presence of bilateral Millers Class I or II gingival recession defects,
* Periodontally healthy patients,
* Patient who demonstrate acceptable oral hygiene status prior to surgical procedure,
* Patient with a medium to deep palatal vault (for Control Group only),
* Patients agreed to give informed consent

Exclusion Criteria:

* History of prolonged use of antibiotics / steroids /immunosuppressive agents/aspirin/anticoagulants/other medications,
* Pregnant women,
* Smokers,
* History of systemic diseases like hypertension, diabetes, HIV, bone metabolic disorders, radiation therapy, immunosuppressive therapy, cancer, etc.
* Patients with unacceptable oral hygiene,
* Faulty tooth brushing technique,
* Mal-aligned tooth,
* Cervical abrasion,
* Teeth with prominent roots.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Reduction in recession depth | Baseline to 6 months
  Recession depth reduction from baseline to 6 months

SECONDARY OUTCOMES:
Reduction in Mean plaque scores | baseline to 6 months
  Mean plaque score reduction form baseline to 6 months
Reduction in mean gingival scores | Baseline to 6 months
  Mean gingival score reduction from baseline to 6 months
Width of keratinised tissue | baseline to 6 months
  Mean keratinised tissue increase from baseline to 6 months
Change Relative attachment level | baseline to 6 months
  Gain in relative attachment level from baseline to 6 months

IPD SHARING:
Plan to Share IPD: No